CLINICAL TRIAL: NCT04494282
Title: The Economic Impact of the Pancreatography in the Endoscopic Treatment of Pancreatic Pseudocysts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Angela Saúl, Principal investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: INCMNSZ
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pseudocyst Pancreas; Pancreatic Duct Disorder
Keywords: Pancreatic Pseudocyst
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Intervention Model Description: Random control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same day (Active Comparator): The ERP will be performed the same day of the endoscopic drainage of PP
  Interventions: Procedure: Endoscopic retrograde pancreatography
- Other day (Active Comparator): The ERP will be performed 6 weeks after the endoscopic drainage of PP.
  Interventions: Procedure: Endoscopic retrograde pancreatography

INTERVENTIONS:
Procedure: Endoscopic retrograde pancreatography — Endoscopic cannulation of main pancreatic duct

SUMMARY:
Pancreatic pseudocysts (PP) present as a complication that occurs in 5-15% of acute pancreatitis and 26-40% of chronic pancreatitis (1-3). To date the endoscopic drainage with endoscopic ultrasound (EUS) has replace the surgical treatment due to the similar success and complication rate but with a lower cost and short hospital stay (4-6). Regarding recurrence, it is important to know the anatomy of the main pancreatic duct (MPD). For this purpose, the endoscopic retrograde pancreatography (ERP) has been describe as a useful tool. In fact, many authors perform it before the endoscopic drainage while others wait several weeks after the drainage (7-9) with similar technical success (5,8). However, there are no studies that compare the technical difficulty and the total cost between these two approaches.

DETAILED DESCRIPTION:
METHODS: Random control trial between two groups. Group 1 the ERP will be performed the same day of the endoscopic drainage of PP. Group 2 the ERP will be performed 6 weeks after the endoscopic drainage of PP. Each ERP will be performed by an expert in ERP in patients who fulfilled the Atlanta criteria for PP. The patients will be enrolled and informed consent will be explained and signed. In those patients who ERP fails, a second attempt will be performed 6 weeks after the endoscopic drainage of PP (Group 1) or a magnetic resonance cholangiopancreatography will be performed (Group 2).

ELIGIBILITY:
Inclusion Criteria:

1. Pancreatic pseudocyst that fulfilled the Atlanta Classification
2. Symptomatic pancreatic pseudocyst
3. Informed consent obtained

Exclusion Criteria:

1. Patient unwilling to participate
2. Absence of duration time of the pancreatography procedure in the record
3. Absence of the number of weeks between the drainage and the pancreatography

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
The impact of the pancreatography in the endoscopic treatment of pancreatic pseudocysts | 6 weeks
  Determine the impact of the timing performing an endoscopic pancreatography in relation of the drainage of pancreatic pseudocyst